CLINICAL TRIAL: NCT02768285
Title: Influence of Maintaining Apical Patency on Postoperative Pain in Posterior Teeth With Necrotic Pulp and Apical Periodontitis: A Randomized Controlled Trial.
Brief Title: Apical Patency and Postoperative Pain.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Isparta Military Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IAH-1
Record Dates: First submitted 2016-05-05; First posted 2016-05-11 (Estimated); Last update posted 2017-10-25 (Actual); Status verified 2016-01

CONDITIONS: Pain Postoperative
Keywords: apical patency; root canal treatment
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention (Experimental): Endodontic treatment was performed in posterior teeth with necrotic pulp and periapical periodontitis using a reciprocating single-file system (Reciproc). Local anesthesia was provided (2% Novocaine with 1:80,000 epinephrine), isolation with rubber dam and standard access cavity preparation was done.Using 2.5 % sodium hypochlorite, canal negotiation was done & apical patency was achieved with #10 K-files in patency group after determining working length. Coronal flaring with # 2 and #3 Gates-Glidden drills was done. The canals were obturated with gutta-percha and epoxy resin sealer. The treatments were carried out in one-visit.
  Interventions: Procedure: APICAL PATENCY
- Control (No Intervention): In the control group, apical patency did not maintained.

INTERVENTIONS:
Procedure: APICAL PATENCY — After determining the working length, a small and flexible size 10 K-file was inserted 1 mm beyond the WL.
  Arms: Intervention

SUMMARY:
The purpose of this study is to determine whether maintaining an apical patency causes postoperative pain in posterior teeth with necrotic pulp and apical periodontitis.

DETAILED DESCRIPTION:
Apical patency (AP) is a procedure that prevents accumulation of soft and hard tissue debris within the cement canal. However, some RCTs indicate that maintaining an AP causes postoperative pain, whilst some RCTs pointed out there is no difference in terms of pain when AP has been performed. We, therefore, would like to conduct a RCT to increase the sample size of the previously performed RCTs to do an systematic review.

ELIGIBILITY:
Inclusion Criteria:

* Mature permanent teeth having plural necrosis and apical periodontitis

Exclusion Criteria:

* Systemic disorders
* Diabetes
* Pregnancy
* Less than 18 years of age
* Immunocompromised
* Patients who had taken antibiotics in the past 1 month
* Patients who had a positive history of analgesic use within the past 3 days
* Previously accessed teeth

Ages: 21 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 320 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2017-07-17 (Actual); Study Completion 2017-08-07 (Actual)

PRIMARY OUTCOMES:
100-mm Visual Analog Scale (VAS). | 7 days.
  Pain severity was evaluated as no pain (0-4 mm), mild pain (5-44 mm), moderate pain (45-74 mm) and severe pain (75-100 mm).

SECONDARY OUTCOMES:
The number of patients taking an analgesic following the endodontic treatment. | 7 days.
  The patients were asked to take an analgesic in the 7 days of time frame.

CONTACTS AND LOCATIONS:
Overall Officials: Ibrahim E YAYLALI, Ph.D., Principal Investigator — Isparta Military Hospital
Locations (1):
- Isparta Military Hospital, Isparta, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes